CLINICAL TRIAL: NCT02641171
Title: Volatiles in Exhaled Breath and Blood in Crohn's Disease: Validation Cohort
Status: Terminated | Type: Observational
Why Stopped: Too slow recruitment and no staff availability
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Agnieszka Smolinska, Postdoc, Maastricht University
Other Study IDs: 00029059
Record Dates: First submitted 2015-12-10; First posted 2015-12-29 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — exhaled air samples blood samples fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Entire Cohort: This is an observational/validation study and there is no intervention involved. Exhaled air samples, blood samples, and fecal samples will be obtained.
  Interventions: Other: Specimen sampling

INTERVENTIONS:
Other: Specimen sampling — exhaled air samples blood samples fecal samples

SUMMARY:
This study evaluates the use of exhaled air analysis as tool to monitor the disease activity in Crohn's Disease (CD). This study is a validation of the previous findings. In this study the participant will be asked to donate exhaled air, blood samples and fecal samples. The breath samples will be used to measure various volatile metabolites in breath. The breath air will be next used to validate the previous findings. The blood samples will be used to define the origin of volatile metabolites in breath. Finally, the potential of exhaled breath analysis as non-invasive marker of diseases activity will be compared to established fecal calprotectin.

DETAILED DESCRIPTION:
In the recent study(doi: 10.1097/Mib.0000000000000436) it was shown the potential of analysis of exhaled air to differentiate active and inactive state of Crohn's Disease (CD). Although, the molecules found in this cohort have shown potential to differentiate between CD patients in remission or with active disease, the validation of the outcomes has to be performed in new population. One crucial pathophysiologic factor in CD is excessive lipid peroxidation during oxidative stress, i.e. during overproduction of oxidants compared to the protective antioxidants. Oxidative stress is a potential aetiological factor and/or a triggering factor in CD. Many volatile compounds including hydrocarbons and aldehydes are produced during oxidative stress and they can be non-invasively measured in exhaled air 5, 6. However, exhaled breath contains volatile metabolites originating from previous or current uptake of environmental contaminants, and more interestingly from metabolism of foreign organisms (bacteria, viruses, fungi or yeasts). Therefore, it is important to study not only exhaled air but also blood in which blood borne volatile molecules can be measured. Since the current study also aims for validating the use of volatile molecules in exhaled air as non-invasive markers for disease activity in CD patients, the investigators will compare the outcome of exhaled air analysis with currently established non-invasive measure of disease activity, i.e. fecal calprotectin.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* BMI: 19-30
* scheduled colonoscopy

Exclusion Criteria:

* disease compromising immune system (such as HIV positive status or patients after organ transplantation
* liver disease
* active and untreated tuberculosis
* chemotherapy agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target population will consist of individuals with established diagnosis of Crohn's Disease (CD). The target population will include male and female between the ages of 18 and 65 years and standard BMI (between 19 and 30). Potential study participants will be excluded if having any disease compromising immune system (such as HIV positive status or patients after organ transplantations), diagnosis of any liver disease, active and untreated tuberculosis and chemotherapy agents. All potential participants must have scheduled appointment for colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds profile: volatile compound concentrations in breath | The samples will be collected within no more than one week before scheduled colonoscopy.
  The exhaled air samples will be used to first validate the volatile compounds for disease activity in Crohn's Disease.
Metabolic profile: metabolite concentrations in blood | The samples will be collected within no more than one week before scheduled colonoscopy.
  Blood samples will be used to better understand the origin of the volatile compounds in breath.
Fecal calprotectin (µg/g) in fecal samples | The samples will be collected within no more than one week before scheduled colonoscopy.
  Fecal calprotectin will be measured as indicator of the migration of neutrophils to the intestinal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Smolinska, PhD, Principal Investigator — Dartmouth/Maastricht University; Corey A Siegel, PhD,MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Smolinska A, Hauschild AC, Fijten RR, Dallinga JW, Baumbach J, van Schooten FJ. Current breathomics--a review on data pre-processing techniques and machine learning in metabolomics breath analysis. J Breath Res. 2014 Jun;8(2):027105. doi: 10.1088/1752-7155/8/2/027105. Epub 2014 Apr 8. PMID 24713999
- [Result] Bodelier AG, Smolinska A, Baranska A, Dallinga JW, Mujagic Z, Vanhees K, van den Heuvel T, Masclee AA, Jonkers D, Pierik MJ, van Schooten FJ. Volatile Organic Compounds in Exhaled Air as Novel Marker for Disease Activity in Crohn's Disease: A Metabolomic Approach. Inflamm Bowel Dis. 2015 Aug;21(8):1776-85. doi: 10.1097/MIB.0000000000000436. PMID 26199990